CLINICAL TRIAL: NCT02896348
Title: Assessment of a Physio-neuro Platform (SynPhNe) for Home-based Retraining of Hand Function in Stroke Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Paolo Bonato, PhD, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-P-000666
Record Dates: First submitted 2016-08-18; First posted 2016-09-12 (Estimated); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Stroke; Hemiparesis
Keywords: Hemiparesis; Stroke; Rehabilitation; Home-based
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- SynPhNe therapy (Experimental): Subjects will be asked to participate in a program of 18 upper-extremity rehabilitation sessions of 60 minutes with SynPhNe platform, over 6 weeks. The sessions will emphasize wrist and fingers movements, including functional activities.
  During week the two first weeks, 6 sessions will be done under therapist supervision at the Motion Analysis Laboratory at Spaulding Rehabilitation Hospital. Over the next 4 to 5 weeks, 10 sessions following exercises prompted by the SynPhNe system will be done unsupervised at home (or under limited supervision at the hospital), 2 sessions will be done at Spaulding Rehabilitation Hospital to review exercises with the SynPhNe system.
  Over the course of the study, participants will wear Axivity sensors to gather information about upper-extremity usage.
  Interventions: Device: SynPhNe platform
- Conventional therapy (Active Comparator): Subjects will be asked to participate in a program of 18 upper-extremity rehabilitation sessions of 60 minutes under therapist supervision over two weeks at the Motion Analysis Laboratory at Spaulding Rehabilitation Hospital. The sessions will emphasize wrist and fingers movements, including functional activities.
  During week the two first weeks, 6 sessions will be done under therapist supervision at the Motion Analysis Laboratory at Spaulding Rehabilitation Hospital. The remaining 10 sessions will be done unsupervised at home, over approximately 4 weeks, and following the therapist home treatment plan. Over that time, 2 visits to Spaulding Rehabilitation will be made to review home treatment plan. Over the course of the study, participants will wear Axivity sensors to gather information about upper-extremity usage.
  Interventions: Other: Conventional therapy

INTERVENTIONS:
Device: SynPhNe platform — SynPhNe is a non-invasive device. It consists of a piece worn around the forearm, a head component and it communicates wirelessly with the computer to provide feedback while performing motor tasks with the hemiparetic hand. The head cap records brain activity and gives feedback to help relaxing while exercising. The arm and the head component communicate wirelessly with the computer via Bluetooth. The head component reads brain signals while the arm gear senses your muscle signals when performing the exercises. The computer software adopts the appropriate difficulty level, speed and duration of the exercise depending on brain and muscle status to minimize fatigue.
  Arms: SynPhNe therapy
Other: Conventional therapy — Exercise program established with a therapist (8 sessions under therapist direct supervision and 10 sessions at home). Low functioning subjects will be given more proximal joint-muscle exercises and activities while higher functioning subjects will have a greater component of distal tasks and activities. The therapist will review the exercises therapy plan with the subject and re-adjust it.
  Arms: Conventional therapy

SUMMARY:
The goal of this study is to:

1. Assess the usability of the SynPhNe device in a home environment.
2. Evaluate the efficacy of the SynPhNe home use device to improve motor hand function in chronic stroke subjects as compared to standard care alone.

DETAILED DESCRIPTION:
The goal of this study is to explore if the SynPhNe system can be used easily at home for people who suffered a stroke. With this study, we are also investigating if the SynPhNe system used could improve your hand function in comparison to conventional therapy.

SynPhNe is a non-invasive device. It consists of a piece worn around the forearm, a head component and it communicates wirelessly via Bluetooth with the computer to provide subject with feedback while performing motor tasks with their hand. The head cap records your brain activity and gives feedback to help relaxing while exercising.

The SynPhNe system has not been approved by the U.S. Food and Drug Administration.

Study participants will be randomized by chance (like a coin toss) to one of the two groups: lab-based upper extremity research therapy or the SynPhNe system for home-based exercises.

* The lab-based upper-extremity research therapy in its content is similar to regular occupational therapy and will focus exercise movements of arm and hand.
* The group testing the SynPhNe system at home will have the system lent at no cost.

The study lasts for up to 12 weeks and involves up to 22 sessions in total:

* Up to 3 sessions will be for testing arm movements (at baseline, after research therapy and at 1 month follow-up).
* 18 research therapy sessions. 10 of them will be done at Spaulding Rehabilitation Hospital with a therapist and 8 of them by yourself, at home. Study participants will either be using the SynPhNe system or the therapy plan recommended by the therapist, depending on the randomization. Each of these visits will be an hour long. They will be scheduled 3 days per week for six weeks.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic or hemorrhagic stroke at least 6 months prior study enrollment ;
* Moderate upper-extremity hemiparesis (initial score on the Upper Extremity Fugl-Meyer Assessment between 21 and 55 out of 66) ;
* Ability to extend at least 2 fingers in the affected hand 10 degrees at any joint with pain-free passive range of motion at least 50% in all joints below the elbow.

Exclusion Criteria:

* Cognitive impairment resulting to inability to follow instructions (as assessed with the MMSE) and inability to sustain attention for more than 10 minutes;
* Current participation in upper-extremity therapy program;
* Treatment with Botox injections in the affected arm in the previous 3 months and no planned Botox injections before the end of the study;
* Aphasia sufficient to limit comprehension and completion of the treatment protocol;
* No more than moderate impairments in paretic UE sensation, passive range of motion, and pain that would limit ability to engage in therapy;
* Increased muscle tone as indicated by score of >/= 3 on the Modified Ashworth Scale;
* Previous diagnosis of dementia;
* Previous diagnosis of neurological diseases other than Stroke;
* History of seizures disorder and/or a seizure occuring within the last 6 months;
* Other conditions affecting function of the stroke affected upper limb;
* Severe pain in the stroke affected upper limb;
* Terminal diseases with expected survival <1 year;

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Upper Extremity - Motor | Week 0, Week 7, Week 11
  This is a motor function assessment for stroke survivors who have hemiplegia. Items are scored on a 3-point ordinal scale where 0=cannot perform, 1=performs partially, and 2=performs fully.
  Higher scores are indicative of higher function. Maximum score=66.
Box and Block Test | Week 0, Week 7, Week 11
  The test is an assessment of unilateral gross manual dexterity. It is performed with each hand separately, the stroke-affected hand and the non-affected hand.
  The scored is calculated by counting the number of blocks that were carried over the partition from one side of the box to the other side of the box in 1 minute. Higher scores are indicative of better gross manual dexterity.
Wolf Motor Function Test - Functional Ablility | Week 0, Week 7, Week 11
  This assessment evaluates motor ability of the upper extremity during timed and functional tasks.
  Functional ability scores are assigned using a 6-point ordinal scale, and the maximum score is 75. A score of 0=does not attempt with the involved arm and a score of 5=arm does participate; movement appears to be normal. Higher scores are indicative of higher function.
Wolf Motor Function Test - Performance Time | Week 0, Week 7, Week 11
  This assessment evaluates motor ability of the upper extremity during timed and functional tasks.
  Performance time is measured in seconds, with up to 120 seconds allowed.

SECONDARY OUTCOMES:
Grip Strength | Week 0, Week 7, Week 11
  This is a measurement of maximal isometric hand grip strength in kilograms. A Jamar dynamometer will be utilized.
Visual Analogue Scale for Pain | Week 0, Week 7, Week 11
  This is an assessment of pain intensity from 0=no pain to 10=worse pain imaginable.
Spasticity -- Modified Ashworth Scale | Week 0, Week 7, Week 11
  The upper extremity will be assessed for spasticity. Scores will be assigned based on the Modified Ashworth Scale. Scores range from from 0=no spasticity/ no increase in muscle tone) to 4=affected part(s) rigid in flexion or extension.
Motor Activity Log - Amount of Use | Week 0, Week 7, Week 11
  This outcome measure assesses upper extremity function and use through patient report.
  Items are scored using a 6-point ordinal scale. For the Amount Scale, 0=the weaker arm was not used at all for that activity (not used), while 5=the weaker arm was used as often as before the stroke (same as pre-stroke).
  The score is calculated by adding the rating scores for each item and dividing by the number of items asked.
EQ5D Questionnaire | Week 0, Week 7, Week 11
  This is a health questionnaire that evaluates quality of life in 5 dimensions including mobility, self-care, usual activities, pain/discomfort, and anxiety/depressions. Applicable to a wide range of health conditions and treatments, the EQ-5D health questionnaire provides a simple descriptive profile and a single index value for health status. Answers are coded as a number where 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=unable or extreme problems.
  An index score is calculated and ranges from 0=a state as bad as being dead to 1=full health.
Motor Activity Log - Quality of Movement | Week 0, Week 7, Week 11
  This outcome measure assesses upper extremity function and use through patient report.
  Items are scored using a 6-point ordinal scale. For the How Well Scale, 0=the weaker arm was not used at all for that activity (not used), while 5=the ability to use the weaker arm for that activity was as good as before the stroke (normal).
  The score is calculated by adding the rating scores for each item and dividing by the number of items asked.

OTHER OUTCOMES:
Range of Motion -- Upper Extremity | Week 0, Week 7, Week 11
  Upper-extremity range of motion is assessed utilizing a goniometer.
Manual Muscle Testing | Week 0, Week 7, Week 11
  This is an assessment of muscle strength. Scores will be assigned according to the Kendall Muscle Strength Grading System. Scores range from 0 (no contraction felt or seen) to 5 (holds test position against strong pressure).
Device Satisfaction Feedback Questionnaire (only for intervention group) | Week 7
  This questionnaire gathers satisfaction feedback about the usage of the device. Questions are scored from 1 to 5, with a total score up to 25. Higher scores indicate higher satisfaction with the device.
Systolic and Diastolic Blood Pressure | Week 0, Week 7, Week 11
  Blood pressure measurement is collected on the non-affected upper limb. Units are mmHg.
Number of Sessions Completed (only for intervention group) | Week 7
  This is a log of completed sessions recorded by the software. Higher numbers indicates better adherence to the intervention.
Number of Issues Encountered with the Device and/or Software (only for intervention group) | Week 7
  This is a recording of the number of occurrences of device and/or software malfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Bonato, PhD, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No